CLINICAL TRIAL: NCT04581148
Title: Determination of SARS-CoV2 Antibody Prevalence in Pediatric Patients
Brief Title: SARS-CoV2 Antibodies in Pediatric Patients (COVID-19)
Acronym: SARS-CoV2_KIDS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: 405_20 Bc
Record Dates: First submitted 2020-10-03; First posted 2020-10-09 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: SARS-Cov2
Keywords: SARS-Cov2; Pediatrics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (10):
- M6: All inpatient and outpatient patients of the Department of Pediatric- and Adolescent medicine of the University Hospital Erlangen in 4 weeks (M6) with residual blood samples.
  Interventions: Diagnostic Test: Blood test antibodies against SARS-CoV-2
- M12: All inpatient and outpatient patients of the Department of Pediatric- and Adolescent medicine of the University Hospital Erlangen in 4 weeks (M12) with residual blood samples.
  Interventions: Diagnostic Test: Blood test antibodies against SARS-CoV-2
- M15: All inpatient and outpatient patients of the Department of Pediatric- and Adolescent medicine of the University Hospital Erlangen in 4 weeks (M15) with residual blood samples.
  Interventions: Diagnostic Test: Blood test antibodies against SARS-CoV-2
- M19: All inpatient and outpatient patients of the Department of Pediatric- and Adolescent medicine of the University Hospital Erlangen in 4 weeks (M19) with residual blood samples.
  Interventions: Diagnostic Test: Blood test antibodies against SARS-CoV-2
- M21: All inpatient and outpatient patients of the Department of Pediatric- and Adolescent medicine of the University Hospital Erlangen in 4 weeks (M21) with residual blood samples.
  Interventions: Diagnostic Test: Blood test antibodies against SARS-CoV-2
- M22: All inpatient and outpatient patients of the Department of Pediatric- and Adolescent medicine of the University Hospital Erlangen in 4 weeks (M22) with residual blood samples.
  Interventions: Diagnostic Test: Blood test antibodies against SARS-CoV-2
- M23: All inpatient and outpatient patients of the Department of Pediatric- and Adolescent medicine of the University Hospital Erlangen in 4 weeks (M23) with residual blood samples.
  Interventions: Diagnostic Test: Blood test antibodies against SARS-CoV-2
- M24: All inpatient and outpatient patients of the Department of Pediatric- and Adolescent medicine of the University Hospital Erlangen in 4 weeks (M24) with residual blood samples.
  Interventions: Diagnostic Test: Blood test antibodies against SARS-CoV-2
- M25: All inpatient and outpatient patients of the Department of Pediatric- and Adolescent medicine of the University Hospital Erlangen in 4 weeks (M25) with residual blood samples.
  Interventions: Diagnostic Test: Blood test antibodies against SARS-CoV-2
- M26: All inpatient and outpatient patients of the Department of Pediatric- and Adolescent medicine of the University Hospital Erlangen in 4 weeks (M26) with residual blood samples.
  Interventions: Diagnostic Test: Blood test antibodies against SARS-CoV-2

INTERVENTIONS:
Diagnostic Test: Blood test antibodies against SARS-CoV-2 — Residual blood of inpatients and outpatients will be analyzed anonymous with a quantitative test for the assessment of antibodies against SARS-CoV-2
  Other Names: Quantitative test for the assessment of antibodies against SARS-CoV-2

SUMMARY:
Since the beginning of the year, the entire world has been concerned with the novel SARS-CoV2 virus. After the first case descriptions in Wuhan, there has been a rapid increase in the number of cases in Germany as well. In case of an illness with the virus, the affected patients can suffer from a slight infection of the upper respiratory tract up to severe lung failure and death. Interestingly, up to now, children are usually less severely affected than adults. However, the actual infection rates are probably similar to those of adults, even if the actual prevalence in children is difficult to quantify so far. The extent of the disease in children has also been less researched to date than in adults, and the same applies to pregnant women and their newborns. In addition, intensive research into possible therapeutic strategies and new vaccines is necessary. Here, however, the number of clinical studies in children is also far behind. In order to be able to understand the infection process and to protect the population with their children, comprehensive testing is necessary. However, this poses great challenges for local health authorities. Scientific investigations are also costly, but are already being carried out by many institutes. So far, for example in the SeBlueCo study, a very low prevalence of antibodies (1.3% of people) has been show. In children, however, both the routes of infection and the way the immune system deals with the virus are probably different than in adults. In this study the investigators now want to examine residual blood samples from pediatric patients of the pediatric and adolescent clinic in the time course after the beginning of the pandemic in order to better understand and monitor the development of antibody prevalence.

DETAILED DESCRIPTION:
Since the beginning of the year, the entire world has been concerned with a novel virus called SARS-CoV2. After the first case descriptions in Wuhan, there has been a rapid increase in the number of cases in Germany as well. In the case of a disease with the virus, the patients affected can suffer from a slight infection of the upper respiratory tract to severe lung failure and death. Since the beginning of the pandemic, an increasing number of complications such as thromboses, kidney failure and neurological damage have also been described. Interestingly, to date, children are usually less severely affected than adults, but the actual infection rates are probably similar to those of adults5 , although the actual prevalence in children is difficult to quantify and has so far been localized. The actual extent of the disease in children has also been little researched to date, and the same applies to pregnant women and their newborns.

In order to be able to understand the course of infection as well as possible and to protect the population, comprehensive testing is necessary. However, this poses great challenges for local health authorities. In addition, intensive research into possible therapy strategies and new vaccines is necessary. Here, however, the number of clinical trials in children is far behind. For adult patients, symptomatic therapies such as immunosuppressive drugs (dexamethasone) and controversially discussed antiviral drugs (e.g. ritonavir) are currently available. The medium-term goal, the establishment of a vaccine, seems to be within reach, but an exact date is not foreseeable.

In the future, in addition to the detection of the active virus by molecular diagnostic tests, the quantitative serological detection of antibodies will also be important in order to be able to make epidemiological statements about herd immunization or vaccination. An interim analysis of the SeBlueCo study showed a proportion of just 1.3% seropositive individuals among blood donors. Similar studies have already been registered and partially conducted throughout Germany. Some studies are also investigating pediatric patients, as both the routes of infection and the way the immune system deals with the virus are probably different from those in adults. Furthermore, the time course of antibody concentrations after infection with SARS-CoV2 and thus the duration of a safe immunity is much discussed. In this study, the investigators want to quantify the prevalence of SARS-Cov2 antibodies in children and adolescents during the pandemic, in order to describe the extent of antibody formation depending on various factors.

At the Children and Youth Clinic Erlangen, at least one blood sample will be taken from all inpatients and most of the patients treated as outpatients. At least one EDTA and one lithium heparin and often also one serum tube is taken. Due to the in-house laboratory, the analysis is designed for very small blood volumes. Therefore there is almost always some residual blood left in the blood tubes, which is then stored for about 7 days and only then discarded (reserve sample). For the study now planned, these residual blood samples from paediatric patients of the paediatric and adolescent clinic will serve as a basis for the analysis. The timing is such that 6, 12, 18 and 24 months after the outbreak of the pandemic in Germany, a SARS-Cov2 antibody prevalence of the local area will be determined. This will allow to investigate the local infection situation as well as the influence of a possibly available vaccination on the extent of immunization in the future.

ELIGIBILITY:
Inclusion Criteria:

* residual blood sample

Exclusion Criteria:

* insufficient blood in the residual blood sample

Ages: 1 Minute to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All patients who were treated in the respective month (M6, M12, M15, M18, M24) in the Department of Children and Adolescent Medicine as outpatients, inpatients or semi-inpatients.
Sampling Method: Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of antibodies against SARS-CoV-2 at timepoint "M6, M12, M15, M19, M21, M22, M23, M24, M25 and M26" | Single assessment per patient in "M6, M12, M15, M19, M21, M22, M23, M24, M25 and M26"
  Prevalence of antibodies against SARS-CoV-2 at timepoint "M6, M12, M15, M19, M21, M22, M23, M24, M25 and M26"

SECONDARY OUTCOMES:
Quantitative antibodies against SARS-CoV-2 at timepoint "M6, M12, M15, M19, M21, M22, M23, M24, M25 and M26" | Single assessment per patient in "M6, M12, M15, M19, M21, M22, M23, M24, M25 and M26"
  Quantitative antibodies against SARS-CoV-2 at timepoint "M6, M12, M15, M19, M21, M22, M23, M24, M25 and M26"
Rate of SARS-CoV-2 antibodies in comparison between month M6, M12, M15, M19, M21, M22, M23, M24, M25 and M26 | Single assessment per patient in "M6, M12, M15, M19, M21, M22, M23, M24, M25 and M26"
  Rate of SARS-CoV-2 antibodies in comparison between month M6, M12, M15, M19, M21, M22, M23, M24, M25 and M26
Stratification of the antibodies against SARS-Cov-2 with patient characteristics (age, gender, clinical history) at timepoint "M6, M12, M15, M19, M21, M22, M23, M24, M25 and M26" | Single assessment per patient in "M6, M12, M15, M19, M21, M22, M23, M24, M25 and M26"
  Stratification of the antibodies against SARS-Cov-2 with patient characteristics (age, gender, clinical history) at timepoint "M6, M12, M15, M19, M21, M22, M23, M24, M25 and M26"

CONTACTS AND LOCATIONS:
Overall Officials: Antje Neubert, PhD, Principal Investigator — Department of Pediatric- and Adolescent Medicine, FAU Erlangen-Nürneberg
Locations (1):
- University Hospital Erlangen, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Dong Y, Mo X, Hu Y, Qi X, Jiang F, Jiang Z, Tong S. Epidemiology of COVID-19 Among Children in China. Pediatrics. 2020 Jun;145(6):e20200702. doi: 10.1542/peds.2020-0702. Epub 2020 Mar 16. PMID 32179660
- [Background] Bhopal SS, Bagaria J, Bhopal R. Risks to children during the covid-19 pandemic: some essential epidemiology. BMJ. 2020 Jun 10;369:m2290. doi: 10.1136/bmj.m2290. No abstract available. PMID 32522815
- [Background] Nicoletti A, Talarico V, Sabetta L, Minchella P, Colosimo M, Fortugno C, Galati MC, Raiola G. Screening of COVID-19 in children admitted to the hospital for acute problems: preliminary data. Acta Biomed. 2020 May 11;91(2):75-79. doi: 10.23750/abm.v91i2.9607. PMID 32420929
- [Background] Bi Q, Wu Y, Mei S, Ye C, Zou X, Zhang Z, Liu X, Wei L, Truelove SA, Zhang T, Gao W, Cheng C, Tang X, Wu X, Wu Y, Sun B, Huang S, Sun Y, Zhang J, Ma T, Lessler J, Feng T. Epidemiology and transmission of COVID-19 in 391 cases and 1286 of their close contacts in Shenzhen, China: a retrospective cohort study. Lancet Infect Dis. 2020 Aug;20(8):911-919. doi: 10.1016/S1473-3099(20)30287-5. Epub 2020 Apr 27. PMID 32353347
- [Background] Diriba K, Awulachew E, Getu E. The effect of coronavirus infection (SARS-CoV-2, MERS-CoV, and SARS-CoV) during pregnancy and the possibility of vertical maternal-fetal transmission: a systematic review and meta-analysis. Eur J Med Res. 2020 Sep 4;25(1):39. doi: 10.1186/s40001-020-00439-w. PMID 32887660
- [Background] Hwang TJ, Randolph AG, Bourgeois FT. Inclusion of Children in Clinical Trials of Treatments for Coronavirus Disease 2019 (COVID-19). JAMA Pediatr. 2020 Sep 1;174(9):825-826. doi: 10.1001/jamapediatrics.2020.1888. No abstract available. PMID 32379296
- [Background] Angus DC, Derde L, Al-Beidh F, Annane D, Arabi Y, Beane A, van Bentum-Puijk W, Berry L, Bhimani Z, Bonten M, Bradbury C, Brunkhorst F, Buxton M, Buzgau A, Cheng AC, de Jong M, Detry M, Estcourt L, Fitzgerald M, Goossens H, Green C, Haniffa R, Higgins AM, Horvat C, Hullegie SJ, Kruger P, Lamontagne F, Lawler PR, Linstrum K, Litton E, Lorenzi E, Marshall J, McAuley D, McGlothin A, McGuinness S, McVerry B, Montgomery S, Mouncey P, Murthy S, Nichol A, Parke R, Parker J, Rowan K, Sanil A, Santos M, Saunders C, Seymour C, Turner A, van de Veerdonk F, Venkatesh B, Zarychanski R, Berry S, Lewis RJ, McArthur C, Webb SA, Gordon AC; Writing Committee for the REMAP-CAP Investigators; Al-Beidh F, Angus D, Annane D, Arabi Y, van Bentum-Puijk W, Berry S, Beane A, Bhimani Z, Bonten M, Bradbury C, Brunkhorst F, Buxton M, Cheng A, De Jong M, Derde L, Estcourt L, Goossens H, Gordon A, Green C, Haniffa R, Lamontagne F, Lawler P, Litton E, Marshall J, McArthur C, McAuley D, McGuinness S, McVerry B, Montgomery S, Mouncey P, Murthy S, Nichol A, Parke R, Rowan K, Seymour C, Turner A, van de Veerdonk F, Webb S, Zarychanski R, Campbell L, Forbes A, Gattas D, Heritier S, Higgins L, Kruger P, Peake S, Presneill J, Seppelt I, Trapani T, Young P, Bagshaw S, Daneman N, Ferguson N, Misak C, Santos M, Hullegie S, Pletz M, Rohde G, Rowan K, Alexander B, Basile K, Girard T, Horvat C, Huang D, Linstrum K, Vates J, Beasley R, Fowler R, McGloughlin S, Morpeth S, Paterson D, Venkatesh B, Uyeki T, Baillie K, Duffy E, Fowler R, Hills T, Orr K, Patanwala A, Tong S, Netea M, Bihari S, Carrier M, Fergusson D, Goligher E, Haidar G, Hunt B, Kumar A, Laffan M, Lawless P, Lother S, McCallum P, Middeldopr S, McQuilten Z, Neal M, Pasi J, Schutgens R, Stanworth S, Turgeon A, Weissman A, Adhikari N, Anstey M, Brant E, de Man A, Lamonagne F, Masse MH, Udy A, Arnold D, Begin P, Charlewood R, Chasse M, Coyne M, Cooper J, Daly J, Gosbell I, Harvala-Simmonds H, Hills T, MacLennan S, Menon D, McDyer J, Pridee N, Roberts D, Shankar-Hari M, Thomas H, Tinmouth A, Triulzi D, Walsh T, Wood E, Calfee C, O'Kane C, Shyamsundar M, Sinha P, Thompson T, Young I, Bihari S, Hodgson C, Laffey J, McAuley D, Orford N, Neto A, Detry M, Fitzgerald M, Lewis R, McGlothlin A, Sanil A, Saunders C, Berry L, Lorenzi E, Miller E, Singh V, Zammit C, van Bentum Puijk W, Bouwman W, Mangindaan Y, Parker L, Peters S, Rietveld I, Raymakers K, Ganpat R, Brillinger N, Markgraf R, Ainscough K, Brickell K, Anjum A, Lane JB, Richards-Belle A, Saull M, Wiley D, Bion J, Connor J, Gates S, Manax V, van der Poll T, Reynolds J, van Beurden M, Effelaar E, Schotsman J, Boyd C, Harland C, Shearer A, Wren J, Clermont G, Garrard W, Kalchthaler K, King A, Ricketts D, Malakoutis S, Marroquin O, Music E, Quinn K, Cate H, Pearson K, Collins J, Hanson J, Williams P, Jackson S, Asghar A, Dyas S, Sutu M, Murphy S, Williamson D, Mguni N, Potter A, Porter D, Goodwin J, Rook C, Harrison S, Williams H, Campbell H, Lomme K, Williamson J, Sheffield J, van't Hoff W, McCracken P, Young M, Board J, Mart E, Knott C, Smith J, Boschert C, Affleck J, Ramanan M, D'Souza R, Pateman K, Shakih A, Cheung W, Kol M, Wong H, Shah A, Wagh A, Simpson J, Duke G, Chan P, Cartner B, Hunter S, Laver R, Shrestha T, Regli A, Pellicano A, McCullough J, Tallott M, Kumar N, Panwar R, Brinkerhoff G, Koppen C, Cazzola F, Brain M, Mineall S, Fischer R, Biradar V, Soar N, White H, Estensen K, Morrison L, Smith J, Cooper M, Health M, Shehabi Y, Al-Bassam W, Hulley A, Whitehead C, Lowrey J, Gresha R, Walsham J, Meyer J, Harward M, Venz E, Williams P, Kurenda C, Smith K, Smith M, Garcia R, Barge D, Byrne D, Byrne K, Driscoll A, Fortune L, Janin P, Yarad E, Hammond N, Bass F, Ashelford A, Waterson S, Wedd S, McNamara R, Buhr H, Coles J, Schweikert S, Wibrow B, Rauniyar R, Myers E, Fysh E, Dawda A, Mevavala B, Litton E, Ferrier J, Nair P, Buscher H, Reynolds C, Santamaria J, Barbazza L, Homes J, Smith R, Murray L, Brailsford J, Forbes L, Maguire T, Mariappa V, Smith J, Simpson S, Maiden M, Bone A, Horton M, Salerno T, Sterba M, Geng W, Depuydt P, De Waele J, De Bus L, Fierens J, Bracke S, Reeve B, Dechert W, Chasse M, Carrier FM, Boumahni D, Benettaib F, Ghamraoui A, Bellemare D, Cloutier E, Francoeur C, Lamontagne F, D'Aragon F, Carbonneau E, Leblond J, Vazquez-Grande G, Marten N, Wilson M, Albert M, Serri K, Cavayas A, Duplaix M, Williams V, Rochwerg B, Karachi T, Oczkowski S, Centofanti J, Millen T, Duan E, Tsang J, Patterson L, English S, Watpool I, Porteous R, Miezitis S, McIntyre L, Brochard L, Burns K, Sandhu G, Khalid I, Binnie A, Powell E, McMillan A, Luk T, Aref N, Andric Z, Cviljevic S, Dimoti R, Zapalac M, Mirkovic G, Barsic B, Kutlesa M, Kotarski V, Vujaklija Brajkovic A, Babel J, Sever H, Dragija L, Kusan I, Vaara S, Pettila L, Heinonen J, Kuitunen A, Karlsson S, Vahtera A, Kiiski H, Ristimaki S, Azaiz A, Charron C, Godement M, Geri G, Vieillard-Baron A, Pourcine F, Monchi M, Luis D, Mercier R, Sagnier A, Verrier N, Caplin C, Siami S, Aparicio C, Vautier S, Jeblaoui A, Fartoukh M, Courtin L, Labbe V, Leparco C, Muller G, Nay MA, Kamel T, Benzekri D, Jacquier S, Mercier E, Chartier D, Salmon C, Dequin P, Schneider F, Morel G, L'Hotellier S, Badie J, Berdaguer FD, Malfroy S, Mezher C, Bourgoin C, Megarbane B, Voicu S, Deye N, Malissin I, Sutterlin L, Guitton C, Darreau C, Landais M, Chudeau N, Robert A, Moine P, Heming N, Maxime V, Bossard I, Nicholier TB, Colin G, Zinzoni V, Maquigneau N, Finn A, Kress G, Hoff U, Friedrich Hinrichs C, Nee J, Pletz M, Hagel S, Ankert J, Kolanos S, Bloos F, Petros S, Pasieka B, Kunz K, Appelt P, Schutze B, Kluge S, Nierhaus A, Jarczak D, Roedl K, Weismann D, Frey A, Klinikum Neukolln V, Reill L, Distler M, Maselli A, Belteczki J, Magyar I, Fazekas A, Kovacs S, Szoke V, Szigligeti G, Leszkoven J, Collins D, Breen P, Frohlich S, Whelan R, McNicholas B, Scully M, Casey S, Kernan M, Doran P, O'Dywer M, Smyth M, Hayes L, Hoiting O, Peters M, Rengers E, Evers M, Prinssen A, Bosch Ziekenhuis J, Simons K, Rozendaal W, Polderman F, de Jager P, Moviat M, Paling A, Salet A, Rademaker E, Peters AL, de Jonge E, Wigbers J, Guilder E, Butler M, Cowdrey KA, Newby L, Chen Y, Simmonds C, McConnochie R, Ritzema Carter J, Henderson S, Van Der Heyden K, Mehrtens J, Williams T, Kazemi A, Song R, Lai V, Girijadevi D, Everitt R, Russell R, Hacking D, Buehner U, Williams E, Browne T, Grimwade K, Goodson J, Keet O, Callender O, Martynoga R, Trask K, Butler A, Schischka L, Young C, Lesona E, Olatunji S, Robertson Y, Jose N, Amaro dos Santos Catorze T, de Lima Pereira TNA, Neves Pessoa LM, Castro Ferreira RM, Pereira Sousa Bastos JM, Aysel Florescu S, Stanciu D, Zaharia MF, Kosa AG, Codreanu D, Marabi Y, Al Qasim E, Moneer Hagazy M, Al Swaidan L, Arishi H, Munoz-Bermudez R, Marin-Corral J, Salazar Degracia A, Parrilla Gomez F, Mateo Lopez MI, Rodriguez Fernandez J, Carcel Fernandez S, Carmona Flores R, Leon Lopez R, de la Fuente Martos C, Allan A, Polgarova P, Farahi N, McWilliam S, Hawcutt D, Rad L, O'Malley L, Whitbread J, Kelsall O, Wild L, Thrush J, Wood H, Austin K, Donnelly A, Kelly M, O'Kane S, McClintock D, Warnock M, Johnston P, Gallagher LJ, Mc Goldrick C, Mc Master M, Strzelecka A, Jha R, Kalogirou M, Ellis C, Krishnamurthy V, Deelchand V, Silversides J, McGuigan P, Ward K, O'Neill A, Finn S, Phillips B, Mullan D, Oritz-Ruiz de Gordoa L, Thomas M, Sweet K, Grimmer L, Johnson R, Pinnell J, Robinson M, Gledhill L, Wood T, Morgan M, Cole J, Hill H, Davies M, Antcliffe D, Templeton M, Rojo R, Coghlan P, Smee J, Mackay E, Cort J, Whileman A, Spencer T, Spittle N, Kasipandian V, Patel A, Allibone S, Genetu RM, Ramali M, Ghosh A, Bamford P, London E, Cawley K, Faulkner M, Jeffrey H, Smith T, Brewer C, Gregory J, Limb J, Cowton A, O'Brien J, Nikitas N, Wells C, Lankester L, Pulletz M, Williams P, Birch J, Wiseman S, Horton S, Alegria A, Turki S, Elsefi T, Crisp N, Allen L, McCullagh I, Robinson P, Hays C, Babio-Galan M, Stevenson H, Khare D, Pinder M, Selvamoni S, Gopinath A, Pugh R, Menzies D, Mackay C, Allan E, Davies G, Puxty K, McCue C, Cathcart S, Hickey N, Ireland J, Yusuff H, Isgro G, Brightling C, Bourne M, Craner M, Watters M, Prout R, Davies L, Pegler S, Kyeremeh L, Arbane G, Wilson K, Gomm L, Francia F, Brett S, Sousa Arias S, Elin Hall R, Budd J, Small C, Birch J, Collins E, Henning J, Bonner S, Hugill K, Cirstea E, Wilkinson D, Karlikowski M, Sutherland H, Wilhelmsen E, Woods J, North J, Sundaran D, Hollos L, Coburn S, Walsh J, Turns M, Hopkins P, Smith J, Noble H, Depante MT, Clarey E, Laha S, Verlander M, Williams A, Huckle A, Hall A, Cooke J, Gardiner-Hill C, Maloney C, Qureshi H, Flint N, Nicholson S, Southin S, Nicholson A, Borgatta B, Turner-Bone I, Reddy A, Wilding L, Chamara Warnapura L, Agno Sathianathan R, Golden D, Hart C, Jones J, Bannard-Smith J, Henry J, Birchall K, Pomeroy F, Quayle R, Makowski A, Misztal B, Ahmed I, KyereDiabour T, Naiker K, Stewart R, Mwaura E, Mew L, Wren L, Willams F, Innes R, Doble P, Hutter J, Shovelton C, Plumb B, Szakmany T, Hamlyn V, Hawkins N, Lewis S, Dell A, Gopal S, Ganguly S, Smallwood A, Harris N, Metherell S, Lazaro JM, Newman T, Fletcher S, Nortje J, Fottrell-Gould D, Randell G, Zaman M, Elmahi E, Jones A, Hall K, Mills G, Ryalls K, Bowler H, Sall J, Bourne R, Borrill Z, Duncan T, Lamb T, Shaw J, Fox C, Moreno Cuesta J, Xavier K, Purohit D, Elhassan M, Bakthavatsalam D, Rowland M, Hutton P, Bashyal A, Davidson N, Hird C, Chhablani M, Phalod G, Kirkby A, Archer S, Netherton K, Reschreiter H, Camsooksai J, Patch S, Jenkins S, Pogson D, Rose S, Daly Z, Brimfield L, Claridge H, Parekh D, Bergin C, Bates M, Dasgin J, McGhee C, Sim M, Hay SK, Henderson S, Phull MK, Zaidi A, Pogreban T, Rosaroso LP, Harvey D, Lowe B, Meredith M, Ryan L, Hormis A, Walker R, Collier D, Kimpton S, Oakley S, Rooney K, Rodden N, Hughes E, Thomson N, McGlynn D, Walden A, Jacques N, Coles H, Tilney E, Vowell E, Schuster-Bruce M, Pitts S, Miln R, Purandare L, Vamplew L, Spivey M, Bean S, Burt K, Moore L, Day C, Gibson C, Gordon E, Zitter L, Keenan S, Baker E, Cherian S, Cutler S, Roynon-Reed A, Harrington K, Raithatha A, Bauchmuller K, Ahmad N, Grecu I, Trodd D, Martin J, Wrey Brown C, Arias AM, Craven T, Hope D, Singleton J, Clark S, Rae N, Welters I, Hamilton DO, Williams K, Waugh V, Shaw D, Puthucheary Z, Martin T, Santos F, Uddin R, Somerville A, Tatham KC, Jhanji S, Black E, Dela Rosa A, Howle R, Tully R, Drummond A, Dearden J, Philbin J, Munt S, Vuylsteke A, Chan C, Victor S, Matsa R, Gellamucho M, Creagh-Brown B, Tooley J, Montague L, De Beaux F, Bullman L, Kersiake I, Demetriou C, Mitchard S, Ramos L, White K, Donnison P, Johns M, Casey R, Mattocks L, Salisbury S, Dark P, Claxton A, McLachlan D, Slevin K, Lee S, Hulme J, Joseph S, Kinney F, Senya HJ, Oborska A, Kayani A, Hadebe B, Orath Prabakaran R, Nichols L, Thomas M, Worner R, Faulkner B, Gendall E, Hayes K, Hamilton-Davies C, Chan C, Mfuko C, Abbass H, Mandadapu V, Leaver S, Forton D, Patel K, Paramasivam E, Powell M, Gould R, Wilby E, Howcroft C, Banach D, Fernandez de Pinedo Artaraz Z, Cabreros L, White I, Croft M, Holland N, Pereira R, Zaki A, Johnson D, Jackson M, Garrard H, Juhaz V, Roy A, Rostron A, Woods L, Cornell S, Pillai S, Harford R, Rees T, Ivatt H, Sundara Raman A, Davey M, Lee K, Barber R, Chablani M, Brohi F, Jagannathan V, Clark M, Purvis S, Wetherill B, Dushianthan A, Cusack R, de Courcy-Golder K, Smith S, Jackson S, Attwood B, Parsons P, Page V, Zhao XB, Oza D, Rhodes J, Anderson T, Morris S, Xia Le Tai C, Thomas A, Keen A, Digby S, Cowley N, Wild L, Southern D, Reddy H, Campbell A, Watkins C, Smuts S, Touma O, Barnes N, Alexander P, Felton T, Ferguson S, Sellers K, Bradley-Potts J, Yates D, Birkinshaw I, Kell K, Marshall N, Carr-Knott L, Summers C. Effect of Hydrocortisone on Mortality and Organ Support in Patients With Severe COVID-19: The REMAP-CAP COVID-19 Corticosteroid Domain Randomized Clinical Trial. JAMA. 2020 Oct 6;324(13):1317-1329. doi: 10.1001/jama.2020.17022. PMID 32876697
- [Background] Beigel JH, Tomashek KM, Dodd LE, Mehta AK, Zingman BS, Kalil AC, Hohmann E, Chu HY, Luetkemeyer A, Kline S, Lopez de Castilla D, Finberg RW, Dierberg K, Tapson V, Hsieh L, Patterson TF, Paredes R, Sweeney DA, Short WR, Touloumi G, Lye DC, Ohmagari N, Oh MD, Ruiz-Palacios GM, Benfield T, Fatkenheuer G, Kortepeter MG, Atmar RL, Creech CB, Lundgren J, Babiker AG, Pett S, Neaton JD, Burgess TH, Bonnett T, Green M, Makowski M, Osinusi A, Nayak S, Lane HC; ACTT-1 Study Group Members. Remdesivir for the Treatment of Covid-19 - Final Report. N Engl J Med. 2020 Nov 5;383(19):1813-1826. doi: 10.1056/NEJMoa2007764. Epub 2020 Oct 8. PMID 32445440
- [Background] Ali MJ, Hanif M, Haider MA, Ahmed MU, Sundas F, Hirani A, Khan IA, Anis K, Karim AH. Treatment Options for COVID-19: A Review. Front Med (Lausanne). 2020 Jul 31;7:480. doi: 10.3389/fmed.2020.00480. eCollection 2020. PMID 32850922
- [Background] Neupane K, Ahmed Z, Pervez H, Ashraf R, Majeed A. Potential Treatment Options for COVID-19: A Comprehensive Review of Global Pharmacological Development Efforts. Cureus. 2020 Jun 26;12(6):e8845. doi: 10.7759/cureus.8845. PMID 32754388
- [Background] Iyer AS, Jones FK, Nodoushani A, Kelly M, Becker M, Slater D, Mills R, Teng E, Kamruzzaman M, Garcia-Beltran WF, Astudillo M, Yang D, Miller TE, Oliver E, Fischinger S, Atyeo C, Iafrate AJ, Calderwood SB, Lauer SA, Yu J, Li Z, Feldman J, Hauser BM, Caradonna TM, Branda JA, Turbett SE, LaRocque RC, Mellon G, Barouch DH, Schmidt AG, Azman AS, Alter G, Ryan ET, Harris JB, Charles RC. Dynamics and significance of the antibody response to SARS-CoV-2 infection. medRxiv [Preprint]. 2020 Jul 20:2020.07.18.20155374. doi: 10.1101/2020.07.18.20155374. PMID 32743600